CLINICAL TRIAL: NCT02274298
Title: Improving Care for Patients With Chronic Kidney Disease Using Electronic Medical Record Interventions: A Pragmatic Cluster Randomized Trial
Brief Title: Improving Care for Patients With Chronic Kidney Disease Using EMRALD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Ontario Renal Network (Unknown)
Responsible Party: Principal Investigator, Dr. Karen Tu, Senior Scientist, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 074-2013-2
Record Dates: First submitted 2014-10-06; First posted 2014-10-24 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CKD feedback and tools (Active Comparator): Physicians in these clinics/clusters will receive feedback on their performance for screening and managing CKD quality indicators as well as EMR tools to aid in their performance
  Interventions: Behavioral: CKD feedback and tools
- No Intervention (No Intervention): Physicians in these clinics/clusters will not receive CKD feedback or tools

INTERVENTIONS:
Behavioral: CKD feedback and tools — people in the intervention arm will receive feedback on ckd quality indicators and tools to help in the detection and management of ckd
  Arms: CKD feedback and tools

SUMMARY:
This pragmatic cluster randomized controlled trial will test the impact of feedback and a toolkit aimed at improving the management of chronic kidney disease (CKD) in the primary care setting. This trial will use family physicians in Ontario participating in the Electronic.

DETAILED DESCRIPTION:
This trial will use family physicians in Ontario participating in the Electronic Medical Record Administrative data Linked Database (EMRALD) and receiving the System for Audit and Feedback to Improve caRE (SAFIRE) along with other decision support tools. Performance on CKD quality indicators for family physicians receiving the CKD feedback and tools will be compared to physicians not receiving the CKD feedback or tools.

ELIGIBILITY:
Inclusion Criteria:

* Family physicians participating in EMRALD, on the EMR for >=2 years, roster size >=100 patients
* Patient criteria, rostered and actively seeing an EMRALD physician, on the EMR for .=1 year

Exclusion Criteria:

* Updated data available at the time of study commencement

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2014-10; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients age 50-80 with Stage 3+ CKD and a statin prescription | 24 months
  Comparison of proportion of patients age 50-80 years with Stage 3+ CKD (no dialysis or renal transplant) and receiving a statin prescription at baseline and at the end of the trial

SECONDARY OUTCOMES:
Proportion of patients at high risk screened for CKD with an eGFR and/or ACR | 24 months
  compare baseline rates to end of intervention rates
Proportion of patients with an initial eGFR <60 and a f/u eGFR or an ACR | 24 months
  compare baseline rates to end of intervention rates
Proportion of patients with diabetes and albuminuria and on an ACE or ARB | 24 months
  compare baseline rates to end of intervention rates
Proportion of patients meeting eGFR criteria for CKD and documentation of CKD in the cumulative patient profile (CPP) | 24 months
  compare baseline rates to end of intervention rates
Proportion of patients with an ACR in the past 18 months and meeting bp targets | 24 months
  compare baseline rates to end of intervention rates
Proportion of patients age less than 80 years and an eGFR<30 being seen by or with a referral to a Nephrologist | 24 months
  compare baseline rates to end of intervention rates

CONTACTS AND LOCATIONS:
Overall Officials: Karen Tu, MD, MSc, Principal Investigator — ICES/Sunnybrook

IPD SHARING:
Plan to Share IPD: No
No, final results will be aggregate although as part of the trial individual participants do receive individual level feedback

REFERENCES:
- [Derived] Nash DM, Ivers NM, Young J, Jaakkimainen RL, Garg AX, Tu K. Improving Care for Patients With or at Risk for Chronic Kidney Disease Using Electronic Medical Record Interventions: A Pragmatic Cluster-Randomized Trial Protocol. Can J Kidney Health Dis. 2017 Apr 5;4:2054358117699833. doi: 10.1177/2054358117699833. eCollection 2017. PMID 28607686